CLINICAL TRIAL: NCT00639665
Title: Cocoa, Polyphenols, and the Kidney in Healthy Subjects and in Subjects With Hypertension and Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: MasterFoods (Industry)
Responsible Party: Principal Investigator, Norman K. Hollenberg, MD, PhD, Director Physiologic Research, Brigham and Women's Hospital
Other Study IDs: 2000P-002347
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
Keywords: Cocoa, diabetes, polyphenols
MeSH Terms: conditions — Diabetes Mellitus | interventions — Chocolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole red blood cells will be retained for DNA analysis. Subjects may "opt-out" of genetic testing.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cocoa — Polyphenol rich or poor cocoa was administered to study subjects to measure hemodynamic responses and the role of nitric oxide in the renal vasodilator response.

SUMMARY:
Observing how cocoa effects the cardiovascular and renal system.

DETAILED DESCRIPTION:
Study designed to assess the vascular benefits of drinking Cocoa that is rich in polyphenols. Vascular beds studied will include kidney, brain, eye, and periphery (finger). Time course of the effects will be studied in healthy normal (including elderly), and also in subjects with Type I and Type II diabetes. Renal blood flow will be determined by PAH/In u test clearance. Cranial ultrasound will be used to measure brain blood flow. Retinal blood flow will be assessed by specialized ultrasound/doppler device. Peripheral blood flow is measured by plethysmography. Urine and blood samples will be assayed for routine physiologic parameters, including hormone assessment, and also for the presence of cocoa metabolites.

ELIGIBILITY:
Inclusion Criteria: Diabetes (Type I and II), with or without Hypertension, blood pressure <165/105

Exclusion Criteria: Under 18 or over 85 years old, women who are pregnant or able to become pregnant, history of heart attack, stroke or chest pain within the past 6 months, kidney disease, heart disease, severe high blood pressure not controlled by medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic (Type I and II)
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Measurements | Hourly measurements (5-6 hours total)

SECONDARY OUTCOMES:
Blood Pressure | Hourly (5-6 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Hollenberg, M.D., Ph.D., Principal Investigator — Brigham and Women's Hospital; Ebrahim Barkouadh, M.D., M.P.H., Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States